CLINICAL TRIAL: NCT06971497
Title: Cleveland Clinic ActivBraid Rotator Cuff Repair (RCR) Study
Brief Title: Zimmer ActivBraid Rotator Cuff Repair (RCR) Study
Status: Recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Principal Investigator, Kathleen Derwin, PhD, Associate Staff Scientist, The Cleveland Clinic
Other Study IDs: 25-252
Record Dates: First submitted 2025-04-29; First posted 2025-05-14 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Rotator Cuff Repair of the Shoulder
Keywords: rotator cuff repair; shoulder; rotator cuff tear; collagen suture
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- patients undergoing primary arthroscopic rotator cuff repair: Patients undergoing primary arthroscopic rotator cuff repair will have their repair completed with ActivBraid™Collagen Co-Braid suture (Zimmer Biomet).
  Interventions: Device: ActivBraid™Collagen Co-Braid suture (Zimmer Biomet)

INTERVENTIONS:
Device: ActivBraid™Collagen Co-Braid suture (Zimmer Biomet) — ActivBraid™ is a suture made from approximately half ultra-high molecular weight polyethylene and and half collagen derived from cow skin. Collagen is the most abundant protein in our bodies and serves as the building block for tendons and bones. The collagen in ActivBraid™ is intended to enhance cell attachment and tissue integration which may improve the healing of a rotator cuff repair. ActivBraid™ suture has been shown to have equivalent strength as other high strength sutures used in orthopaedic procedures and has been approved by the Food and Drug Administration (FDA) for repairing tendons. ActivBraid™ is a commercially available product that has been and is used in humans. This is the first post-market clinical study with ActivBraid™.

SUMMARY:
We will enroll up to 65 patients undergoing primary arthroscopic rotator cuff repair (RCR) using ActivBraid™Collagen Co-Braid suture (Zimmer Biomet) and evaluate RCR healing as well as shoulder range of motion, strength, and patient-reported outcomes at 6m, 1y and 2y.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years
* acute or chronic, reparable, 1-5 cm full thickness tear of the supraspinatus and/or infraspinatus tendons

Exclusion Criteria:

* prior ipsilateral shoulder surgery
* outstanding worker's compensation claim
* symptomatic cervical spine disease
* a frozen shoulder
* advanced glenohumeral arthritis
* isolated subscapularis tear
* significant radiation exposure for other medical reasons.
* known is advance to be claustrophobic
* known history of hypersensitivity to bovine-derived materials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing primary arthroscopic rotator cuff repair
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Rotator cuff repair healing | 1 year post-operation
  Patients will undergo magnetic resonance imaging (MRI) of the shoulder from which healing of their rotator cuff repair will be classified using Sugaya score from 1-5, where higher score indicated worse healing.
Rotator cuff repair healing | 1 year post-operation
  Patients will also undergo computed tomography (CT) scans of the shoulder from which tendon retraction of the rotator cuff repair will also be measured in millimeters where higher tendon retraction indicates worse healing.

SECONDARY OUTCOMES:
Patient-reported outcome measures | 1 year post-operation
  Patients will be asked to answer the American Shoulder and Elbow Surgeons (ASES) Score from 0-100 points where higher score indicates better outcome.
Shoulder strength | 1 year post-operation
  Isometric shoulder strength in pounds will be assessed using a table mounted dynamometer.
Shoulder range of motion | 1 year post-operation
  Shoulder range-of-motion will be assessed by asking patients to lift their affected arm overhead in the scapular plane and measuring the range with a manual goniometer (degrees).

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Derwin, PhD, Principal Investigator — The Cleveland Clinic; Eric Ricchetti, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: product information for ActivBraid™Collagen Co-Braid suture (Zimmer Biomet) — https://www.zimmerbiomet.com/en/products-and-solutions/specialties/sports-medicine/activbraid.html